CLINICAL TRIAL: NCT07247552
Title: Personalized Pain Treatment by Transcranial Magnetic Stimulation in Patients With Chronic Pain: A Prospective Interventional Study With Embedded Predictive Biomarker Evaluation
Brief Title: Personalized Treatment by rTMS in Chronic Pain - Study2
Acronym: PersoNINpain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Margit Midtgaard Bach, Dr., Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20230076-3
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
Keywords: Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Chronic Pain; Transcranial Magnetic Stimulation; Neuromodulation
MeSH Terms: conditions — Chronic Pain; Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms

STUDY DESIGN:
Masking Description: Patients and investigators are blinded to the prediction of whether a participant is expected to become a responder or non-responder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Classical rTMS to M1 (Active Comparator): This is a prospective, single-arm interventional study designed to evaluate the predictive value of a neurophysiological biomarker for rTMS response in chronic pain patients. Patients will be allocated to two groups according to their baseline M1 connectivity at baseline in a 1:1 proportion. Patients with "low" connectivity will be compared to controls having "high" connectivity. All patients will receive repetitive transcranial magnetic stimulation (rTMS) to the primary cortex (M1). Low connectivity will be defined by TMS-EEG evoked responses. Responses to a single pulse of TMS delivered to M1 before therapy. TMS-EEG responses will be analysed by phase- and power-based metrics such as global mean field power and inter-trial coherence in the alpha band, according to previous studies. The study main hypothesis is that pre-therapy M1 low connectivity is a predictor of response to M1 rTMS.
  Interventions: Device: rTMS to M1

INTERVENTIONS:
Device: rTMS to M1 — • The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds with an interval of twenty seconds between trains will be delivered, as traditionally performed. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes. All patients will receive 14 sessions of rTMS.

SUMMARY:
Previous research has shown the effectiveness of magnetic stimulation of the brain as a supplemental treatment for various conditions, such as depression and chronic pain. However, the application of magnetic stimulation has been standardized across patients without considering individual differences. This one-size-fits-all approach results in only half of the patients benefiting from the treatment, with the other half seeing no improvement in their symptoms. Therefore, a study on individuals with chronic pain will be performed to explore how magnetic stimulation treatments can be tailored to each person. This will involve analysing brain signal measurements before the start of the therapy and adjusting/personalizing the magnetic stimulations to each individual person.

DETAILED DESCRIPTION:
This is a prospective, single-arm interventional study designed to evaluate the predictive value of a neurophysiological biomarker for repetitive transcranial magnetic stimulation (rTMS) response in chronic pain patients. The project aims to test if the effects of non-pharmacological, non-invasive pain treatment can be enhanced by employing brain connectivity information to guide the application of rTMS. Previous efficacy and safety trials have supported that current best practice for rTMS for pain relief in chronic pain patients, is applied to one cortical area: primary motor cortex (M1). However, only around 50% respond to the treatment. Since there is no current strategy to know which patient will respond to treatment, patients with chronic pain end up undergoing trial and error strategies, which delay their improvement. This is actually not different from challenges related to pharmacological treatment, where each medication only relieves pain in 30-40% of patients, and the choice of each medication is based on "trial-and-error basis".

Several strategies currently aim to provide a more individualized strategy for choosing analgesic interventions based on patient-related information. To allow for the design of efficacy trials in the future, the present project is based on a proof-of-concept, mechanistic design. It will employ M1 rTMS stimulation for pain reduction. However, based on everyone's brain signals as read by EEG recorded before the start of the treatment it will be determined whether the patient is most likely to respond or not. Therefore, before receiving a full rTMS treatment, patients will undergo a neurophysiological screening session using single-pulse TMS-EEG. Single-pulse TMS and EEG have been routinely used in the clinic as a part of the neurophysiological assessment of patients for decades but have not yet been used in the association as an attempt to try to guide who will become a responder to the treatment. In the screening session, single pulses TMS will be applied to the primary network hub used as current best-practice in therapeutic rTMS: M1. Concomitantly, the EEG oscillatory activity of this cortical area will be recorded, and the brain connectivity state will be assessed. By using information derived from a patient´s brain connectivity state using transcranial magnetic stimulation with electroencephalography (TMS-EEG), it will be determined if the participant is most likely to respond or not. High oscillatory activity is expected to result in becoming a non-responder.

A total of 90 subjects with chronic pain will be included in a double-blind, randomized two parallel-arm study aiming to be able to accurately predict who will become a responder and a non-responder based on high oscillatory activity.

In the initial baseline measurement, the subjects will fill out questionnaires and undergo neurophysiological assessments which include rest EEG, TMS-EEG of M1, rTMS-EEG, followed by a repetition of TMS-EEG of M1 and rest EEG. After this baseline measurement, the subjects will receive daily rTMS sessions targeting M1 (called induction phase) for 5 consecutive days (Monday to Friday). Each of the 5 daily stimulations will last 30 minutes, of which 15 minutes will be under treatment.

The induction phase will be followed by a 7-week maintenance phase, with 1 rTMS session per week (totalling 7 rTMS sessions). At the end of the maintenance phase, primary and secondary outcomes (questionnaires) will be collected to investigate the efficacy of the rTMS treatments. These questionnaires will also be sent to participants 12 weeks following end of treatment. A random subsample of 30 participants will be asked if they would like to participate in a second 3-hour neurophysiological assessment to investigate the changes in brain connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic pain (present most of the days for more than 3 months).
* Pain with a mean pain intensity between 3-9 on a 0-10 pain scale (where 0 means no pain and 10 means the worst pain imaginable).
* Speak and understand English or Danish

Exclusion Criteria:

* Pregnant or breastfeeding
* Current uncontrolled major depression as the main diagnosis
* Current history of substance abuse
* Lack of ability to cooperate, to fully understand the protocol or any difficulty in filling out questionnaires (e.g., due to language or cognitive problems)
* Formal contraindications to TMS application (presence of epilepsy, cranial implanted ferromagnetic devices, e.g., intracranial neurostimulator or cochlear implants, tattoos with metal ink on the face or permanent make up with metal in the face )
* Unable to answer the "Transcranial Magnetic Stimulation Adult Safety Screen" screening questionnaire.
* Participation in other research protocols within 1 month before the inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual analogue scale) | VAS will be assessed before treatment and post intervention. Responders are those with ≥30% pain reduction, based on the difference in VAS the last 24 hours at the end of maintenance compared to average pain intensity the week before baseline assessment.
  The '0' represents 'no pain' at all, and '100' represents the 'worst possible pain' that the individual can imagine.

SECONDARY OUTCOMES:
Patients' Global Impression of Change | Patients' Global Impression of Change will be investigated before the treatment, at the end of the course of treatment (8 weeks of treatment), and again after 3 months following the end of treatment.
  The questionnaire assesses the individual's impression of change after an intervention.
  The Likert scale is asking whether 'After the beginning of this study, my overall state of health is': with the options of 'Very much improved', 'Much improved', 'Minimally improved', 'No change', 'Minimally worse', 'Much worse'.
Short Brief Pain Inventory | Short Brief Pain Inventory changes will be investigated before the treatment, at the end of the course of treatment (8 weeks of treatment), and again after 3 months following the end of treatment.
  9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Items such as pain severity and Pain Interference Score can be calculated as well as number of affected body areas.
Short McGill Pain Questionnaire | Short McGill Pain Questionnaire changes will be investigated before the treatment, at the end of the course of treatment (8 weeks of treatment), and again after 3 months following the end of treatment.
  A comprehensive multidimensional tool that assesses the three main aspects of pain: sensory discriminative, affective-motivational, and cognitive-evaluative. Words describing pain is presented and the patient has to choose whether it is recognisable in mild, moderate or severe way and it has the option of 'none'.
Quality of sleep (VAS) | Sleep VAS changes will be investigated before the treatment, at the end of the course of treatment (8 weeks of treatment), and again after 3 months following the end of treatment.
  A VAS scale to determine 'how did you sleep last night' ranging from 0 ('poor') to 10 ('great').

CONTACTS AND LOCATIONS:
Overall Officials: Margit M Bach, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No